CLINICAL TRIAL: NCT03807388
Title: The Use of ReMindCare Application for Smartphone in Treatment of Patients From First Episode of Psychosis Unit in the Clinic Hospital of Valencia, Spain.
Brief Title: ReMindCare App for Patients From First Episode of Psychosis Unit.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigacion Sanitaria INCLIVA (Other)
Collaborators: University of Valencia (Other); Universitat Politècnica de València (Other); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Lucia Bonet, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/059
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Psychosis; Schizophrenia; Psychotic Disorders; Delirium; Hallucinations; Adherence, Medication; Treatment Side Effects
Keywords: eHealth; mHealth; smartphone; app; psychosis; adherence; early intervention
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Delirium; Hallucinations; Medication Adherence; Alzheimer Disease | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ReMindCare Intervention Group (Experimental): Patients from First Episode of Psychosis Unit who will use ReMindCare app.
  ReMindCare is an user-friendly app which conducts daily evaluations of the health status of patients with psychosis by some quick questions that patients will have to answer.
  Interventions: Device: ReMindCare Intervention Group
- Treatment as Usual (Other): Patients from First Episode of Psychosis Unit who will follow psychiatric usual care.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Device: ReMindCare Intervention Group — Daily and weekly assessments of patient´s health status, and generation of alarms related to these answers. Moreover, patients can contact clinicians by an urgent consultation tab.
  Other Names: ReMindCare app
  Arms: ReMindCare Intervention Group
Other: Treatment as Usual — Psychiatric usual treatment at First Episode of Psychosis Unit at Clinical Hospital of Valencia, Spain.
  Arms: Treatment as Usual

SUMMARY:
ReMindCare is an app designed by the Unit of Psychiatry at the Clinical Hospital of Valencia in liaison with the Polytechnic University of Valencia.

This e-Health app gathers information about the clinical health status of patients with Psychotic Disorder Diagnose through daily and weekly brief assessments.

This information is displayed in a restricted access website, where clinicians can visualize data from patients as well as download pdf reports of main data collected by the app. These reports can be attached to the electronic clinical report of the patient at the hospital database, being accessible for consultation for every clinician involved in treatment of the patient.

Furthermore, ReMindCare produces different alarms which notify clinicians about variations into patients health status or the cessation of using the app. Moreover, patients can also deliberately generate an urgent consultation alarm.

The introduction of ReMindCare app into clinical practice will follow a clinical trial structure in which treatment as usual (TAU) of patients from a First Episode of Psychosis Unit will be compared to ReMindCare app intervention program. After participants eligible for inclusion complete baseline assessments they will be randomly allocated to one of the two groups (Intervention or TAU) by a basic single blind randomization in which an independent researcher will perform the allocation using a computerized random number generator.

Information collected through the app and variations into clinical data will be analyzed among time. First assessment of these data will be conducted after 6 months of patient´s enrollment into the study. Subsequent analysis will be conducted yearly.

DETAILED DESCRIPTION:
Baseline surveys:

Baseline surveys will be administered. In this first evaluation, sociodemographic information and clinical information such as diagnosis, pattern of antipsychotic treatment, number of suicide attempts or associated illnesses will be collected.

Furthermore, some structured questionnaires will be administered, including: Clinical Global Impression Scale (CGI), Global Assessment of Functioning (GAF), Positive and Negative Syndrome Scale (PANSS), Premorbid Adjustment Scale (PAS), Simplified Medication Adherence Questionnaire (SMAQ), Drug Attitude Inventory (DAI-10) and Beck Cognitive Insight Scale (BCIS).

ReMindCare app measures:

Patients will generate the following data by using the app:

1. Data generated through responses to daily and weekly app questionnaires: Answers to these questionnaires are presented following a Likert scale (1 to 5) as follows: 1=Not at all, 2=Slightly, 3=Somewhat, 4=Very, 5=Extremely. Responses will be collected and analyzed.
2. Quantity of "Urgent clinic consultation" request made for every patient.
3. Quantity of automatic usage alarms.

Treatment measures:

Apart from data collected through the use of the app, further information will be collected related to modifications into de patient´s treatment or related to his/her health status:

* Modifications into antipsychotic treatment.
* Number of relapses
* Number of visits to hospital urgent care unit.
* Number of hospital admissions

Follow-up measures and satisfaction questionnaire:

Information collected through the app and variations into clinical data will be analyzed among time. First assessment of these data will be conducted after 6 months of patient´s enrollment into the study. Subsequent analysis will be conducted yearly.

Patients will also complete a satisfaction questionnaire after one year using the ReMindCare app or before discontinuing the use the app (if this happens before the first year of use of the app has come). This app feedback questionnaire is made for the purpose of this research and it is based in some previous satisfaction and usability questionnaires such as: User Version of the mobile application rating scale (uMars), System Usability Scale (SUS), EnLight: Tool for mobile and web-based eHealth interventions and App Quality Evaluation (AQEL).

ELIGIBILITY:
Inclusion Criteria:

* Patients from the FEPU at Clinic Hospital of Valencia.
* Diagnosis of Psychotic Disorder following DSMI-5 [32] criteria.
* Age between 17 to 65 years old.
* Owning a smartphone which allows the correct installation and functioning of the App.
* Owning a smartphone which allows internet connection (not necessary permanent)

Exclusion Criteria:

* Severe Mental Disability
* Lack of abilities in using and mastering mobile devices and internet.
* Not to sign informed consent sheet.
* Level of Spanish not fluid.
* Do not have an own smartphone.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Adherence to anti-psychotic treatment | Yearly, up to 2 years
  Adherence to anti-psychotic medication intake. Measured by: Simplified Medication Adherence Questionnaire (SMAQ).
Adherence to treatment | Yearly, up to 2 years
  Number of hospital admissions and urgent care visits
Early relapse detection | Yearly, up to 2 years
  Changes in detection of relapses into psychotic sympthoms. Measured by number of contacts to patients in response to alerts generated by the app.

SECONDARY OUTCOMES:
Alliance between patient and clinician | Yearly, up to 2 years
  Changes in feelings of alliance between patient and clinician. Measured by a Satisfaction Questionnaire, made for the purpose of this research.
Feeling of empowerment related to illness self-management | Yearly, up to 2 years
  Changes in patient´s feelings of empowerment related to illness self-management. Measured by a Satisfaction Questionnaire, made for the purpose of this research.
Changes in comunication between clinicians | Yearly, up to 2 years
  Study of changes related to comunication between clinicians about treatment of patients. Measured qualitatively by a focus group session.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Sanjuán, Study Director — Instituto de Investigacion Sanitaria INCLIVA
Locations (1):
- INCLIVA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the following IPD data. However they will be analyzed as a group:
  Responses to the following questionnaires:
  * Clinical Global Impression Scale (CGI)
  * Global Assessment of Functioning (GAF)
  * Positive and Negative Syndrome Scale (PANSS)
  * Simplified Medication Adherence Questionnaire (SMAQ)
  * Drug Attitude Inventory (DAI-10)
  * Beck Cognitive Insight Scale (BCIS)
  Socio-demographics information such as: Age, gender, ethnicity education, marital status, living situation.
  Answers of patient to ReMindCare app assessments: Daily / weekly responses and alarms generated
  Treatment related measures:
  * Modifications into antipsychotic treatment.
  * Number of relapses
  * Number of visits to hospital urgent care unit.
  * Number of hospital admissions
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data has been sent for publication in an open access journal.

REFERENCES:
- [Background] Bonet L, Izquierdo C, Escarti MJ, Sancho JV, Arce D, Blanquer I, Sanjuan J. Use of mobile technologies in patients with psychosis: A systematic review. Rev Psiquiatr Salud Ment. 2017 Jul-Sep;10(3):168-178. doi: 10.1016/j.rpsm.2017.01.003. Epub 2017 Mar 1. English, Spanish. PMID 28258835
- [Background] Bonet L, Llacer B, Hernandez-Viadel M, Arce D, Blanquer I, Canete C, Escarti M, Gonzalez-Pinto AM, Sanjuan J. Differences in the Use and Opinions About New eHealth Technologies Among Patients With Psychosis: Structured Questionnaire. JMIR Ment Health. 2018 Jul 25;5(3):e51. doi: 10.2196/mental.9950. PMID 30045835